CLINICAL TRIAL: NCT01002014
Title: Preservation of the Nipple Areolar Complex With Skin Sparing Mastectomy
Brief Title: Nipple Sparing Mastectomy - Cosmetic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI NAC-SSM
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Breast Reconstruction; Cosmesis
Keywords: Breast Cancer; Skin Sparing Mastectomy; Breast Cancer Prophylaxis; Nipple Sparing Mastectomy; Nipple Areolar Complex; Mastectomy; Breast Reconstruction; Local recurrence following nipple sparing mastectomy; Cosmetic outcomes following nipple sparing mastectomy; Complications following nipple sparing mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nipple Sparing Mastectomy (Experimental): Patients who undergo nipple sparing mastectomy with preservation of the nipple areolar complex.
  Interventions: Procedure: Nipple Sparing Mastectomy

INTERVENTIONS:
Procedure: Nipple Sparing Mastectomy — Skin sparing mastectomy with preservation of the nipple areolar complex

SUMMARY:
The purpose of this study is to observe the cosmetic outcomes, patient satisfaction, and complications after skin sparing mastectomy with preservation of the nipple areolar complex.

DETAILED DESCRIPTION:
The outcomes will be observed in patients with both known cancer diagnosis and in those with indications for prophylactic mastectomy. The cosmetic appearance and complications will be followed through several post operative visits throughout the duration of the study. This study is conducted in conjunction with the plastic and reconstructive surgeons who will be performing the breast reconstruction procedures. Patient satisfaction will be measured via survey format. In addition, local recurrence rates will be compared to patients undergoing traditional mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mastectomy for cancer and/or prophylaxis
* Age greater than or equal to 18 at time of surgery
* BMI less than or equal to 35
* If mastectomy is indicated for removal of breast cancer, tumor is clinically T1 or T2

Exclusion Criteria:

* Currently smoking
* Prior radiation to the affected breast
* Systemic lupus erythematosus
* Central tumor location and/or tumor within 2 cm of NAC
* Paget's disease of the nipple
* Clinical evidence of tumor involvement in the nipple
* Clinical evidence of axillary nodal tumor involvement
* Lymphovascular invasion of the tumor on core biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-01-21 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Cosmetic Appearance | First Post Operative year
Patient Satisfaction | First Post Operative Year
Presence of tumor in nipple areolar complex frozen section | Duration of Study
Presence of tumor in nipple areolar complex permanent histology | Duration of study

SECONDARY OUTCOMES:
Complications | First Post Operative year
Local Recurrence | One year

CONTACTS AND LOCATIONS:
Overall Officials: Richard L White, MD, Principal Investigator — Carolinas Healthcare
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Vlajcic Z, Zic R, Stanec S, Lambasa S, Petrovecki M, Stanec Z. Nipple-areola complex preservation: predictive factors of neoplastic nipple-areola complex invasion. Ann Plast Surg. 2005 Sep;55(3):240-4. doi: 10.1097/01.sap.0000171680.49971.85. PMID 16106159
- [Background] Crowe JP, Patrick RJ, Yetman RJ, Djohan R. Nipple-sparing mastectomy update: one hundred forty-nine procedures and clinical outcomes. Arch Surg. 2008 Nov;143(11):1106-10; discussion 1110. doi: 10.1001/archsurg.143.11.1106. PMID 19015470
- [Background] Crowe JP Jr, Kim JA, Yetman R, Banbury J, Patrick RJ, Baynes D. Nipple-sparing mastectomy: technique and results of 54 procedures. Arch Surg. 2004 Feb;139(2):148-50. doi: 10.1001/archsurg.139.2.148. PMID 14769571
- [Background] Sacchini V, Pinotti JA, Barros AC, Luini A, Pluchinotta A, Pinotti M, Boratto MG, Ricci MD, Ruiz CA, Nisida AC, Veronesi P, Petit J, Arnone P, Bassi F, Disa JJ, Garcia-Etienne CA, Borgen PI. Nipple-sparing mastectomy for breast cancer and risk reduction: oncologic or technical problem? J Am Coll Surg. 2006 Nov;203(5):704-14. doi: 10.1016/j.jamcollsurg.2006.07.015. Epub 2006 Sep 11. PMID 17084333
- [Background] Stolier AJ, Sullivan SK, Dellacroce FJ. Technical considerations in nipple-sparing mastectomy: 82 consecutive cases without necrosis. Ann Surg Oncol. 2008 May;15(5):1341-7. doi: 10.1245/s10434-007-9753-5. Epub 2008 Feb 7. PMID 18256883
- [Background] Wijayanayagam A, Kumar AS, Foster RD, Esserman LJ. Optimizing the total skin-sparing mastectomy. Arch Surg. 2008 Jan;143(1):38-45; discussion 45. doi: 10.1001/archsurg.143.1.38. PMID 18209151
- [Background] Banerjee A, Gupta S, Bhattacharya N. Preservation of nipple-areola complex in breast cancer--a clinicopathological assessment. J Plast Reconstr Aesthet Surg. 2008 Oct;61(10):1195-8. doi: 10.1016/j.bjps.2007.08.005. Epub 2007 Sep 27. PMID 17901007
- [Background] Loewen MJ, Jennings JA, Sherman SR, Slaikeu J, Ebrom PA, Davis AT, Fitzgerald TL. Mammographic distance as a predictor of nipple-areola complex involvement in breast cancer. Am J Surg. 2008 Mar;195(3):391-4; discussion 394-5. doi: 10.1016/j.amjsurg.2007.12.020. PMID 18207131
- [Background] Laronga C, Kemp B, Johnston D, Robb GL, Singletary SE. The incidence of occult nipple-areola complex involvement in breast cancer patients receiving a skin-sparing mastectomy. Ann Surg Oncol. 1999 Sep;6(6):609-13. doi: 10.1007/s10434-999-0609-z. PMID 10493632
- [Background] Gerber B, Krause A, Reimer T, Muller H, Kuchenmeister I, Makovitzky J, Kundt G, Friese K. Skin-sparing mastectomy with conservation of the nipple-areola complex and autologous reconstruction is an oncologically safe procedure. Ann Surg. 2003 Jul;238(1):120-7. doi: 10.1097/01.SLA.0000077922.38307.cd. PMID 12832974
- [Background] Fitzal F. Can nipple-sparing mastectomy and immediate breast reconstruction with modified extended latissimus dorsi muscular flap improve the cosmetic and functional outcome of patients with breast cancer? World J Surg. 2008 Mar;32(3):499; author reply 500-1. doi: 10.1007/s00268-007-9268-z. No abstract available. PMID 17952495
- [Background] Carlson GW, Losken A, Moore B, Thornton J, Elliott M, Bolitho G, Denson DD. Results of immediate breast reconstruction after skin-sparing mastectomy. Ann Plast Surg. 2001 Mar;46(3):222-8. doi: 10.1097/00000637-200103000-00003. PMID 11293510
- [Background] Lowery JC, Wilkins EG, Kuzon WM, Davis JA. Evaluations of aesthetic results in breast reconstruction: an analysis of reliability. Ann Plast Surg. 1996 Jun;36(6):601-6; discussion 607. doi: 10.1097/00000637-199606000-00007. PMID 8792969